CLINICAL TRIAL: NCT02678832
Title: Social Cognitions and Norms Towards Physical Exercise Among Cancer Patients and Health Care Professionals
Brief Title: Momentum Project Heidelberg - Dealing Actively With a Cancerous Disease
Status: Completed | Type: Observational
Sponsor: Heidelberg University (Other)
Collaborators: German Cancer Research Center (Other); University of Heidelberg Medical Center (Other); National Center for Tumor Diseases, Heidelberg (Other); German Cancer Aid (Other)
Responsible Party: Principal Investigator, Nadine Ungar, Dr., Heidelberg University
Other Study IDs: 110512/111223
Record Dates: First submitted 2016-01-25; First posted 2016-02-10 (Estimated); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Colorectal Cancer; Breast Cancer; Prostate Cancer; Physicians; Nurses
MeSH Terms: conditions — Colorectal Neoplasms; Breast Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Cancer patients: breast cancer prostate cancer colorectal cancer
- Physicians: working in in- and outpatient care
- Oncology nurses: working in in- and outpatient care

SUMMARY:
The study, investigates the current physical activity promotion practices among physicians and nurses, as well as social norms toward physical activity during treatment among cancer patients and among physicians and nurses who treat or counsel cancer patients.

DETAILED DESCRIPTION:
For this purpose, four large surveys with health care professionals (specialized practitioners, N=300; general practitioners, N=300; oncology nurses, N=300) and cancer patients (N=1200, 400 patients each with breast, prostate or colorectal cancer) with a cross-sectional research design are conducted.

Additionally, a follow-up-study with a sub-sample of cancer patients (N=180) will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* HCP are eligible if they meet the following inclusion criteria: Working as an oncological nurse, general practitioner or physician specialized in oncology, radiology, surgery, gynecology, urology, gastroenterology or rehabilitation Signed informed consent
* Patients are eligible if they meet the following inclusion criteria: Patients with a diagnosis of primary tumor or recurrence no longer than 2 years ago who are undergoing chemo- or radiotherapy currently or in the last 2 years Patients undergoing chemo- or radiotherapy currently or no longer than 2 years ago At least 18 years of age Sufficient German language skills Signed informed consent

Exclusion Criteria:

* HCP will be excluded from the trial if they meet the following exclusion criteria: No regular contact with cancer patients
* Patients will be excluded from the trial if they meet the following exclusion criteria: Presence of comorbidities that preclude involvement in exercise programs (e.g. severe pain, advanced heart failure [≥ NYHA III]) Mentally retarded Reduced standing ability and no ability to walk

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Cross-sectional surveys:
  1. 300 specialized practitioners who treat patients with breast, prostate or colorectal cancer (gynecologists, radiologists, urologists, gastroenterologists, oncologists, surgeons)
  2. 300 general practitioners
  3. 50 rehabilitation physicians
  4. 300 oncology nurses
  5. 1200 cancer patients with breast, prostate or colorectal cancer before or during cancer therapy (pre-treatment and primary cancer treatment time period according to PA and Cancer Control (PACC) framework)
  6. Longitudinal follow-up study: 180 patients [sub-sample of (5)] who are recruited before the initiation or at the beginning of their primary cancer treatment
Sampling Method: Non-Probability Sample
Enrollment: 2200 (Actual)
Dates: Start 2015-12; Primary Completion 2018-06 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Social norms and cognitions toward self-management strategies of cancer patients as assessed by the variables of the theory of planned behavior (TPB) | one-time self-report of current cognitions
  Questionnaire items were developed in a pilot study according to the guidelines for a TPB questionnaire described by Ajzen (2006)

SECONDARY OUTCOMES:
Physical activity as assessed with SQUASH | one-time retrospective self-report about the past month
  self-reported physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Monika Sieverding, Prof. Dr., Principal Investigator — Heidelberg University; Karen Steindorf, Prof. Dr., Principal Investigator — German Cancer Research Center (DKFZ) & National Center for Tumor Diseases (NCT), Heidelberg; Joachim Wiskemann, Dr., Principal Investigator — University of Heidelberg Medical Center & National Center for Tumor Diseases (NCT), Heidelberg

REFERENCES:
- [Derived] Haussmann A, Ungar N, Tsiouris A, Schmidt L, Wiskemann J, Steindorf K, Sieverding M. Better not resting: Carving out attitudes and their associations with physical activity in people with cancer. Eur J Cancer Care (Engl). 2022 Sep;31(5):e13622. doi: 10.1111/ecc.13622. Epub 2022 May 22. PMID 35599349
- [Derived] Depenbusch J, Wiskemann J, Haussmann A, Tsiouris A, Schmidt L, Ungar N, Sieverding M, Steindorf K. Impact and Determinants of Structural Barriers on Physical Activity in People with Cancer. Int J Behav Med. 2022 Jun;29(3):308-320. doi: 10.1007/s12529-021-10014-0. Epub 2021 Sep 22. PMID 34550527
- See also: Homepage of the Study — http://www.momentum-projekt.de